CLINICAL TRIAL: NCT01246596
Title: Chronic Presence of Epstein Barr Virus in Epithelial Cells From Gingiva is Associated With Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 10-AOI-01
Record Dates: First submitted 2010-11-17; First posted 2010-11-23 (Estimated); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Chronic Periodontitis; Aggressive Periodontitis; Presence / Absence of EBV
MeSH Terms: conditions — Chronic Periodontitis; Aggressive Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- chronic periodontitis (Active Comparator)
  Interventions: Procedure: dental root planing
- aggressive periodontitis (Active Comparator)
  Interventions: Procedure: dental root planing
- healthy patient (orthodontics extraction) (Active Comparator)
  Interventions: Procedure: dental root planing

INTERVENTIONS:
Procedure: dental root planing — The objective of root planing, otherwise known as conventional periodontal therapy, non-surgical periodontal therapy, or dental prophylaxis is to remove or eliminate the etiologic agents which cause inflammation: dental plaque, its products and calculus,[1] thus helping to establish a periodontium that is free of disease.[2]
  Arms: chronic periodontitis
Procedure: dental root planing — The objective of root planing, otherwise known as conventional periodontal therapy, non-surgical periodontal therapy, or dental prophylaxis is to remove or eliminate the etiologic agents which cause inflammation: dental plaque, its products and calculus, thus helping to establish a periodontium that is free of disease.
  Arms: aggressive periodontitis
Procedure: dental root planing — The objective of root planing, otherwise known as conventional periodontal therapy, non-surgical periodontal therapy, or dental prophylaxis is to remove or eliminate the etiologic agents which cause inflammation: dental plaque, its products and calculus, thus helping to establish a periodontium that is free of disease.
  Arms: healthy patient (orthodontics extraction)

SUMMARY:
The etiopathogenesis of periodontal disease results from complex interaction between infectious agents, mainly including bacteria, and host cellular and humoral immune responses. However it is thought that bacteria-induced pathogenesis is not sufficient alone to explain all biological and clinical features of the destructive periodontal disease. The main hypothesis is that herpesviruses, such as Epstein-Barr Virus, may participate as well by altering epithelial gingival cell biology and consequently may promote the initiation and progression of periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* 10 patients affected by chronic periodontitis
* 10 patients affected by aggressive periodontitis
* 10 healthy patients (orthodontics extraction)
* Subject who have read and understood the information note relative under investigation and who have signed the informed consent
* major patient

Exclusion Criteria:

* Patient with no contre-indication to periodontal treatment
* Patient with serious blood disease
* Patient who exhibits systemic condition incompatible with realization of the study
* Patient treated with oral retinoids, bisphosphonates, oral anticoagulants and anticonvulsivants
* Patient who presents a buccal carcinoma treated with radiotherapy
* Patient who have received during the past 6 months: anti-inflammatory drugs, anti-cancerous or immunosuppressive chemiotherapy
* Patient who presents a linguistic or psychic incapacity to understand information

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2011-01; Primary Completion 2014-05-05 (Actual); Study Completion 2014-05-05 (Actual)

PRIMARY OUTCOMES:
Percentage of gingival epithelial cells infected by EBV (by immunofluorescence and In situ Hybridization) | at time=0

SECONDARY OUTCOMES:
Epithelial tissue infected by EBV (by immunofluorescence and in situ hybridization) | at time = 0
Presence / absence of latency and / or lytic proteins (by immunofluorescence and in situ hybridization) | at time = 0

CONTACTS AND LOCATIONS:
Overall Officials: Severine VINCENT, PH, Principal Investigator — CHU de Nice Hôpital Saint Roch
Locations (1):
- Dr Severine VINCENT, Nice, France